CLINICAL TRIAL: NCT06729125
Title: Posture Stability and Functional Activity Changes After Transcranial Photobiomodulation for Patients With Parkinson's Disease: A Randomized Controlled Trial
Brief Title: Transcranial Photobiomodulation With Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Hosny M Battesha, associate professor hanan hosny M Battesha, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PD , LASER
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: transcranial photobiomodulation, posture instability, Parkinson's disease, modified Parkinson activity scale, Biodex balance system
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental)
  Interventions: Device: transcranial photobiomodulation
- control group (Active Comparator)
  Interventions: Other: exercises training

INTERVENTIONS:
Device: transcranial photobiomodulation — Single-session transcranial laser stimulation was administered with a continuous-wave, 1,064-nm laser (Model CG-5000 Laser, Cell Gen Therapeutics LLC, Dallas, TX).
  Arms: study group
Other: exercises training — balance exercises and others
  Arms: control group

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder after Alzheimer's disease. It is a progressive and disabling disease with significative impact on quality of life. Since it has no cure, available treatment is targeted to improve the symptoms due to a lack of dopamine in the central nervous system. The aim of the study was to see how transcranial photobiomodulation (tPBM) helped patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD,
* Hoehn & Yahr stage I-IV,
* independent gait with or without technical assistance
* stable parkinsonian medication for at least a month before the study star.

Exclusion Criteria:

* comorbidities that affect balance or walking,
* other neurological pathologies besides PD,
* chronic diseases not medically controlled and participation in another physiotherapy program or sport activity during the intervention period or in the month before starting the study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
posture stability | 8 weeks
  The Biodex Balance System (Biodex Medical Systems Inc, USA) Will be used to assess the limit of stability (overall, forward and backward) pre- and post-treatment.

SECONDARY OUTCOMES:
functional activity | 8 weeks
  The modified Parkinson activity scale (mPAS) consist of 14 items arranged on to three domains: chair transfer (2 items), gait akinesia (6 items) and bed mobility (6 items)

CONTACTS AND LOCATIONS:
Locations (1):
- Al Zaytoonah University, Amaan, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33894193/